CLINICAL TRIAL: NCT06251518
Title: Investigating the Effectiveness of Vimida, a Digital Intervention for People Suffering From Post-viral Chronic Fatigue After COVID-19 Infection
Brief Title: Investigating the Effectiveness of Vimida
Acronym: InvidiCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: Medical School Hamburg (Other); Institut Long-Covid Rostock (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vimida RCT 2024
Record Dates: First submitted 2024-01-24; First posted 2024-02-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Long COVID; Post COVID-19 Condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vimida + TAU (Experimental): Participants allocated to the intervention group will receive access to vimida in addition to treatment as usual (TAU).
  vimida is a digital health application designed for individuals with post-Covid conditions who suffer from fatigue, accessible through a web browser. The application focuses on treatment methods derived from cognitive behavioral therapy (CBT). Topics addressed by vimida are psychoeducation, activity and recovery, attention, stress management, sleep management, cognitive restructuring, and social resources.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivational text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 180 days.
  Interventions: Behavioral: vimida
- TAU (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: vimida — Participants will receive access to the digital health intervention vimida in addition to TAU.
  Arms: vimida + TAU

SUMMARY:
This randomized controlled trial (RCT) with 160 patients suffering from fatigue after COVID-19 infection aims to investigate the effectiveness of the unguided digital therapeutic vimida for reducing post-COVID-19 fatigue. Inclusion criteria are: male, female or non-binary, age ≥18 years, diagnosis of post-COVID-19 fatigue, ≥3 months since the last infection with COVID-19, fatigue severity score (cut-off) of ≥ 16 on the Chalder Fatigue Scale (CFQ-11), consent to participation, and sufficient German language skills. Exclusion criteria are a known psychiatric or somatic condition that can explain the fatigue and current participation in a multidisciplinary rehabilitation program aimed to ameliorate the consequences of COVID-19.

Patients will be randomized and allocated to either an intervention group, in which they will receive access to vimida in addition to treatment as usual (TAU; n=80), or to a control group, in which they will receive access to TAU only (n=80).

The primary endpoint will be fatigue symptoms with three months post-allocation (T1) being the primary time point for assessment of effectiveness. Six months post-allocation (T2) will be used as follow-up assessment of endpoints. Secondary endpoints will be depressive symptoms, mental health-related quality of life, work/social functioning, somatic symptoms, and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* male, female or non-binary
* age ≥ 18
* diagnosis of post-COVID-19 fatigue (ICD-10 U08.9, or U09.9 in conjunction with G93.3), secured via a telemedical visit
* ≥ 3 months since COVID-19 infection that preceded fatigue symptoms
* elevated levels of fatigue: cut-off of ≥ 16 on the CFQ-11
* consent to participation
* sufficient knowledge of the German language

Exclusion Criteria:

* known somatic or psychiatric condition that can explain the fatigue (e.g., cancer, multiple sclerosis, severe depression)
* current participation in a multidisciplinary rehabilitation program aimed at ameliorating the consequences of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue symptom severity | 3 months
  Chalder Fatigue Scale (CFQ-11). Total score ranging from 0-33; higher scores mean higher fatigue symptoms (worse outcome).

SECONDARY OUTCOMES:
Depressive symptoms | 3 months
  Patient Health Questionnaire - 9 item version (PHQ-9). Total score ranging from 0-27; higher scores mean higher depressive symptoms (worse outcome).
Health-related quality of life | 3 months
  Assessment of Quality of Life - 8 Dimensions (AQoL-8D). Total score ranging from 0-100; higher scores mean higher quality of life (better outcome).
Functioning | 3 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Somatic symptoms | 3 months
  Patient Health Questionnaire - 15 item version (PHQ-15). Total score ranging from 0-30; higher scores mean higher somatic symptoms (worse outcome).
Anxiety | 3 months
  Generalized Anxiety Disorder Assessment (GAD-7). Total score ranging from 0-21; higher scores mean higher anxiety symptoms (worse outcome).

OTHER OUTCOMES:
Fatigue symptom severity | 6 months
  Chalder Fatigue Scale (CFQ-11). Total score ranging from 0-33; higher scores mean higher fatigue symptoms (worse outcome).
Depressive symptoms | 6 months
  Patient Health Questionnaire - 9 item version (PHQ-9). Total score ranging from 0-27; higher scores mean higher depressive symptoms (worse outcome).
Health-related quality of life | 6 months
  Assessment of Quality of Life - 8 Dimensions (AQoL-8D). Total score ranging from 0-100; higher scores mean higher quality of life (better outcome).
Functioning | 6 months
  Work and Social Adjustment Scale (WSAS). Total score ranging from 0-40; higher scores mean higher impairment (worse outcome).
Somatic symptoms | 6 months
  Patient Health Questionnaire - 15 item version (PHQ-15). Total score ranging from 0-30; higher scores mean higher somatic symptoms (worse outcome).
Anxiety | 6 months
  Generalized Anxiety Disorder Assessment (GAD-7). Total score ranging from 0-21; higher scores mean higher anxiety symptoms (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Schröder, PhD, Principal Investigator — Medical School Hamburg
Locations (1):
- GAIA, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No